CLINICAL TRIAL: NCT05672004
Title: Implementation of the Combined Lifestyle Intervention ProMuscle for Community-living Older Adults in Community-care Practices.
Brief Title: Implementation of ProMuscle in Daily Practice
Acronym: PUMP-fit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: Regiodeal Foodvalley (Unknown)
Responsible Party: Principal Investigator, Patricia van der Laag, Principal investigator, MSc, UMC Utrecht
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: 22/050
Record Dates: First submitted 2022-12-19; First posted 2023-01-05 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Sarcopenia; Frailty; Aging Problems
Keywords: implementation; lifestyle intervention; prevention
MeSH Terms: conditions — Sarcopenia; Frailty

STUDY DESIGN:
Intervention Model Description: stepped wedge cluster trial and mixed methods process analysis
Masking Description: Recipients of ProMuscle are not the target group within this study. Healthcare professionals are the participants of the study, they know that they received the implementation toolbox once they switched to the intervention group
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Implementation as usual (Active Comparator): Healthcare professionals will be instructed to implement ProMuscle in their practice as usual
  Interventions: Other: Implementation as usual
- PUMP-fit strategy: Implementation toolbox (Experimental): Healthcare professionals receive a personal implementation toolbox, tailored to their contexts' barriers for implementation
  Interventions: Other: PUMP-fit strategy (implementation toolbox)

INTERVENTIONS:
Other: PUMP-fit strategy (implementation toolbox) — Healthcare professionals will receive the ProMuscle training from one of the researchers during a one-hour online meeting (during the control period).
  Healthcare professionals will be informed about the platform and toolbox. Healthcare professionals receive a personal log-in for the online platform. Healthcare professionals receive a questionnaire about their readiness for implementation. The results of this questionnaire are directly visible on the platform Within the separate environment of the online platform, healthcare professionals can access their implementation toolbox. The toolbox is tailored to their personal context based on the results of the 'Readinesstool'.
  Arms: PUMP-fit strategy: Implementation toolbox
Other: Implementation as usual — First, healthcare professionals will receive the ProMuscle training from one of the researchers during a one-hour online meeting.
  At the end of the training healthcare professionals are informed about the mandatory conditions to implement ProMuscle (champion, material, approval of management).
  Healthcare professionals receive a questionnaire about their readiness for implementation. The results of this questionnaire are directly visible. Results contain a graph of possible barriers for implementation in their practice.
  Hereafter they will be instructed to start with implementation as usual.
  Arms: Implementation as usual

SUMMARY:
Implementation of a previously shown (cost-)effective combined lifestyle intervention for community living older adults, ProMuscle, in at least four of the eight communities of the 'Foodvalley' in the Netherlands.

DETAILED DESCRIPTION:
ProMuscle is a combined lifestyle intervention that has been shown effective in improving muscle mass, muscle strength, and physical functioning in community-dwelling older adults. Potentially, it could facilitate older people in maintaining their functional independence.

Despite the promising results, ProMuscle is still not part of daily care. Previously factors influencing successful implementation were identified and implementation strategies targeting these factors were developed and formatted as an implementation toolbox for healthcare professionals.

To increase the likelihood of successful implementation of ProMuscle, this study aims to investigate the PUMP-fit strategy (implementation toolbox) effectiveness on the adoption of ProMuscle in community-care

A hybrid type 3 stepped wedge cluster trial with a mixed method analysis will be conducted to assess the effectiveness of the PUMP-fit implementation toolbox. A stepped wedge trail is chosen because of the ability to compare between clusters, but also within clusters.

Moreover, ProMuscle is already found effective, and the researchers hypothesized that the implementation toolbox should be assessable for all healthcare professionals in the 'Foodvalley'. At last, a stepped wedge design is recommended if there is limited time and a small sample of professionals to recruit from in comparison to the total sample size that is needed to detect any effect.

In addition, the researchers hypothesized that the program would be adapted to specific contexts' outcomes from the recipients of ProMuscle will be collected. A hybrid type three trial aims to investigate the implementation as a primary outcome and the effect of the (adapted) intervention as a secondary outcome.

ELIGIBILITY:
To be eligible to participate in this study, healthcare professionals must met the following criteria:

* Physical therapist, lifestyle coach or dietician in one of the communities in the Foodvalley in the Netherlands
* Interested in combined lifestyle programs for older adults
* Frequently involved in maintaining physical functioning in older adults

In and exclusion criteria for older residents receiving ProMuscle are:

Inclusion criteria:

* Aged 65 years or older
* Living in one of the eight communities of the 'Foodvalley' (Ede, Wageningen, Nijkerk, Rhenen, Veenendaal, Barneveld, Scherpenzeel, Renswoude)
* Able to understand Dutch
* Are pre-frail or frail (score 1 or more points on the Fried frailty criteria), or report loss of muscle strength

Exclusion criteria:

- One or more red flags for participating in progressive resistance exercise without consent of a medical specialist or general practitioner

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2024-03-01 (Actual); Study Completion 2024-05-01 (Actual)

PRIMARY OUTCOMES:
Adoption of ProMuscle | 36 weeks
  The number of healthcare professionals delivering ProMuscle is measured with administrative data and the REport of Sustainment Scale (PRESS). Because it is not possible to measure adoption at baseline, The Measure of Innovation-Specific Implementation Intentions (MISII) questionnaire will be used to measure adoptability (the attention to adopt an EBP) at T0
Fidelity of ProMuscle | 36 weeks
  Fidelity is the degree to which an intervention was implemented as prescribed. The number of activities described in the ProMuscle guideline executed by the healthcare professionals will be assessed with a self-report checklist based on the content of the ProMuscle intervention. Comparing the outcomes of fidelity before and after receiving the PUMP-fit strategy can indicate whether the toolbox contributed to the fidelity of delivery of ProMuscle.

SECONDARY OUTCOMES:
Fidelity of the PUMP-fit strategy | 24 weeks
  Fidelity is the degree to which an intervention was implemented as prescribed. For the PUMP-fit strategy, fidelity is defined as the degree to which the activities described in the online implementation toolbox are implemented as prescribed.
  The number of implementation activities described in the implementation toolbox and the time healthcare professionals are active in the implementation toolbox will be collected from the online platform (tracking activity).
  Fidelity according to healthcare professionals will be assessed with a self-report containing statements based on the Fidelity of Implementation (FOI) framework. The statements are scored with a 5-point Likert scale, the higher the score, the higher the fidelity.
  In addition, the experience of healthcare professionals about the fidelity will be investigated during the process evaluation guided by the domain "implementation" of the RE-AIM framework.
Acceptability of the PUMP-fit strategy | 36 weeks
  Acceptability will be measured with the translated Acceptability of Intervention Measure (AIM). The AIM contains four statements about the acceptability of the PUMP-fit implementation strategy. Statements are scored on a five-point Likert scale. The higher the score the higher the acceptability of the PUMP-fit strategy.
Appropriateness of the PUMP-fit strategy | 36 weeks
  Appropriateness will be measured with the translated Intervention Appropriateness Measure (IAM). The IAM contains four statements about the appropriateness of the PUMP-fit implementation strategy. Statements are scored on a five-point Likert scale. The higher the score the higher the appropriateness of the PUMP-fit strategy.
Feasibility of the PUMP-fit strategy | 36 weeks
  Feasibility will be measured with the translated Feasibility of Intervention Measure (FIM) questionnaire. The FIM contains four statements about the feasibility of the PUMP-fit implementation strategy. Statements are scored on a five-point Likert scale. The higher the score the higher the feasibility of the PUMP-fit strategy.
Barriers and facilitators for implementation of ProMuscle | 36 weeks
  Barriers and facilitators will be assessed with a questionnaire developed by the research group. The questionnaire contains statements about different factors that could influence implementation (CFIR framework) and is based on the 'Wandersman readiness thinking tool' and 'Organization Readiness'. Statements are rated on a 5-point Likert scale. Factors that are scored three or lower will be defined as barriers. Factors that are scored with four of higher will be defined as facilitators.
  Moreover, during the washout period and process evaluation barriers and facilitators will be identified in interviews with healthcare professionals implementing ProMuscle.
Acceptability of ProMuscle | 36 weeks
  Acceptability of ProMuscle will be measured with the translated Acceptability of Intervention Measure (AIM) by the start of the implementation of ProMuscle (T0). Four statements are scored on a five-point Likert scale. The higher the score, the higher the score the higher the acceptability of the ProMuscle intervention
Appropriateness of ProMuscle | 36 weeks
  Appropriateness will be measured with the translated Intervention Appropriateness Measure (IAM) by the start of the implementation of ProMuscle (T0). Four statements are scored on a five-point Likert scale, the higher the score the higher the appropriateness of ProMuscle.
Feasibility of ProMuscle | 36 weeks
  Feasibility will be measured with the translated Feasibility of Intervention Measure (FIM) questionnaire by the start of the implementation of ProMuscle (T0). Four statements are scored on a five-point Likert scale, the higher the score, the higher the score the higher the feasibility of the ProMuscle intervention
Reach of ProMuscle | 36 weeks
  Reach is defined as the number of older adults and will be measured by administrative data.
Sustainment of ProMuscle | 54 weeks
  Sustainment of the implementation of ProMuscle will be measured with the Program Sustainability Assessment Tool (PSAT) and during a one-hour focus group guided by the RE-AIM framework (domain Maintenance) to assess if ProMuscle became part of daily care.
Physical functioning recipients of ProMuscle | 54 weeks
  The Short Physical Performance Battery (SPPB) is conducted by participating healthcare professionals to asses physical functioning.
Functional lower extremity strength recipients of ProMuscle | 54 weeks
  Repeated chair-rise test is conducted by participating healthcare professionals to assess functional strength.
Leg strength recipients of ProMuscle | 54 weeks
  The one repetition (1RM) of leg strength is performed on leg press machines. The 1RM is conducted by participating healthcare professionals.
  The 1RM measures the maximal strength and can be used to develop the exercise program.
Functional mobility recipients of ProMuscle 1RM | 54 weeks
  Functional mobility is measured with the Timed-Up-And-Go test (TUG).
Care dependency recipients of ProMuscle | 54 weeks
  Healthcare professionals report the current health status of the recipients in terms of care dependency. Recipients are asked if they receive care. Answers can be categorized as no care, care from spouse or family, domestic worker, home care, nursing or other help.
Lean body mass recipients ProMuscle | 54 weeks
  Lean body mass is measured with the bioelectrical impedance analysis (BIA)

CONTACTS AND LOCATIONS:
Overall Officials: Lisette Schoonhoven, prof, Principal Investigator — Julius Center, University Medical Center Utrecht, The Netherlands
Locations (1):
- University Medical Center Utrecht, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: No